CLINICAL TRIAL: NCT05916573
Title: A Study to Evaluate the Pharmacokinetics of HSK16149 in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK16149-104
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2022-10

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mild Renal Impairment (Experimental)
  Interventions: Drug: HSK16149
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: HSK16149
- Severe Renal Impairment (Experimental)
  Interventions: Drug: HSK16149
- Normal Renal function (Experimental)
  Interventions: Drug: HSK16149

INTERVENTIONS:
Drug: HSK16149 — single oral adminiatration, 20mg

SUMMARY:
This is an open-label, single-dose study to evaluate the pharmacokinetics and safety of HSK16149 in subjects with mild, moderate and severe renal impairment compared to the matched control subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with renal impairment(RI):

  1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
  2. 18 years to 75 years (inclusive), male and female;
  3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height2 (m^2));
  4. Subjects with medically stable RI until study completion corresponding to the classifications of Renal Function based on GFR: mild RI: 60≤GFR<90 mL/min; moderate RI: 30≤GFR<60 mL/min, severe RI:15≤GFR<30 mL/min;
  5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests results were deemed appropriate by the investigator;
  6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for RI/ other comorbidities (last more than four weeks in good compliance);
  7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration.
* Subjects with normal renal function :

  1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
  2. 18 years to 75 years (inclusive), male and female, age and sex must be matched with subjects with RI;
  3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg, weight must be matched with subjects with RI. Body mass index (BMI) : 18-30 kg/m^2 (inclusive) (BMI= weight (kg)/height2 (m^2));
  4. 90≤GFR<130 mL/min;
  5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests results were deemed appropriate by the investigator;
  6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for comorbidities (last more than four weeks in good compliance);
  7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration.

Exclusion Criteria:

1. Allergic to any component in HSK16149 capsules;
2. Uncontrolled or unstable cardiovascular, respiratory, liver, gastrointestinal tract, endocrine, blood, mental/nervous, etc.Systemic diseases;
3. Those who have committed suicide or suicidal tendency in the past, or those who have recurrent dizziness, headache, memory and cognitive impairment;
4. According to the researcher's judgment, there are factors that affect the absorption, distribution, metabolism and excretion of drugs, such as diseases, drugs, surgery, etc.; Taking Niaoduqing granules, the stool is irregular or shapeless;
5. Acute renal failure;
6. Smoking more than 5 cigarettes a day on average in the 3 months before screening or unable to stop using any tobacco products during the test period;
7. Drinking more than 14 units per week within 3 months before screening (1 unit = 17.7 mL ethanol, that is, 1 unit =357 mL beer with 5% alcohol content, 43 mL white wine with 40% alcohol content or 147 mL wine with 12% alcohol content), or those who can't ban alcohol during the test, or those who are positive in alcohol breath test;
8. Have a history of drug abuse within 5 years before screening, or have a positive drug abuse screening;
9. Those who have ingested beverages or foods rich in xanthine (coffee, tea, chocolate, etc.) or grapefruit for a long time in the past, or have taken any products rich in xanthine or grapefruit orally within 48 hours before administration;
10. Those who have participated in any clinical trials of drugs or medical devices within 3 months before screening (subject to administration).
11. The amount of blood donation (or blood loss) within 3 months before screening is ≥400 mL, or those who have received blood products to improve anemia;
12. One of ALT and/or AST >2*ULN, total bilirubin > 1.5* ULN and creatine kinase > 2*ULN during screening;
13. Those who are positive for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody and treponema pallidum antibody;
14. Female subjects who are pregnant or lactating or whose serum pregnancy results are positive during the screening period or during the trial;
15. Subjects considered by the researcher to have any factors that are not suitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Cmax | From the start to 72 hours after administration
  The maximun plasma concentration of HSK16149
AUC0-t | From the start to 72 hours after administration
  Area under the concentration-time curve from time zero to time of last quantifiable concentration
AUC0-inf | From the start to 72 hours after administration
  Area under the concentration-time curve from time zero extrapolated to infinite time

SECONDARY OUTCOMES:
Tmax | From the start to 72 hours after administration
  Time of maximum concentration
t1/2 | From the start to 72 hours after administration
  half-life
CL | From the start to 72 hours after administration
  Plasma clearance
Vz | From the start to 72 hours after administration
  Volume of distribution associated with the terminal phase
Ae | From the start to 72 hours after administration
  Cumulative urinary recovery of unchanged drug
Fe | From the start to 72 hours after administration
  Cumulative urinary recovery fraction of unchanged drug
CLr | From the start to 72 hours after administration
  Renal clearance

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China